CLINICAL TRIAL: NCT04205981
Title: The Effect of Aerobic Exercise on Body Composition, Cardiovascular System and Autonomic Stress Response, and Cognition in Overweight and Obese Women
Brief Title: The Effect of Aerobic Exercise in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU-2
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Exercise intervention. The experimental group increased their energy expenditure according to American College of Sports Medicine and WHO-based physical activity recommendations for all adults to promote clinically significant weight loss and for additional health benefits: 300 min of moderate-intensity aerobic training throughout the week (WHO, 2010; Swift et al. 2014). Participants underwent five 60 min moderate-intensity cycling sessions per week for a period of 8 weeks, 40 sessions in total. Each session involved 5 min of warm up at 40 Watts, cycling for 50 min at a speed that increased their HR to a target HR obtained at 50-60% of peak VO2, and a 5 min of cool down at 40 Watts.
  Interventions: Other: Aerobic exercise
- Control (No Intervention): . In the control group, participants did not undergo any intervention and were instructed to maintain their regular physical activity and diet regime for 8 weeks.

INTERVENTIONS:
Other: Aerobic exercise — 8-week aerobic exercise (moderate intensity), 5 times per week, 60 min per session. Exercise training under supervision of trained staff.
  Arms: Aerobic exercise

SUMMARY:
Study design The study was designed as a prospective controlled randomized trial. Participants were randomly assigned to one of two groups. In the experimental group, participants (n = 17) received 8-week aerobic exercise intervention without nutrition modifications. In the control group, participants (n = 16) did not undergo any intervention and were instructed to maintain their regular physical activity and diet regime for 8 weeks.

Experimental measurements: Anthropometric measurements, Measurement of BDNF, Cardiac autonomic responses, Measurement of aerobic fitness, Measurement of cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

1. obese women (BMI) > 25 kg/m2;
2. exhibiting weight stability (body weight change < 2 kg) for at least 2 months prior to enrollment;
3. with a sedentary lifestyle (regular exercise < 1 h/week);
4. had no medical condition that would affect study results and limit physical activity;
5. not undergoing lactation;
6. who were not pregnant or postmenopausal.

Ages: 38 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Weight | 8 weeks
  weight (TBF-300 body composition scale; Tanita, UK Ltd., UK) was measured while the participants wore only underwear and were barefoot.
Blood brain-derived neurotrophic factor (BDNF) | 8 weeks
  Venous blood samples (5 mL) were collected and allowed to clot at room temperature. Serum was then separated by centrifugation for 15 min at 1,200 g (room temperature) and stored at -80°C until analysis. BDNF were measured using an enzyme-linked immunoassay system (Gemini; Stratec Biomedical, Birkenfeld, Germany).
Cognitive performance | 8 weeks
  Automated Neuropsychological Assessment Metrics Version 4 (ANAM-4; Vista Life, USA) was used to measure neurocognitive skills: motor reaction time, mental flexibility, mathematical processing, working memory, visual scanning and associative learning skills. Participants were familiarized with the test battery twice before the experiments.
Maximal oxygen uptake | 8 weeks
  Aerobic fitness was assessed by a graded exercise test on an electronically braked cycle ergometer (Ergoselect 100, Ergoline, Bitz, Germany). Standardized verbal encouragement was provided throughout the test to stimulate maximal performance.
Waist and hip circumference | 8 weeks
  Waist circumference was measured to the nearest 0.1 cm, in duplicate, at the level of the iliac crest at the end of the normal expiration. Hip circumference was measured at the maximum protuberance of the buttocks. Waist and hip circumferences were measured at the nearest 0.5 cm.
Resting blood pressure | 8 weeks
  was measured using a digital electronic blood pressure monitor (Microlife BP A100, Widnau, Switzerland)
Heart rate variability | 8 weeks
  R-R intervals were recorded using a Polar H7 sensor with a chest strap (Kempele, Finland).

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No